CLINICAL TRIAL: NCT04271332
Title: An Exploratory, Randomized, Double-Blind, Placebo-Controlled and Open-label Extension Study of the Safety, Tolerability, and Efficacy of Arbaclofen in Subjects With 16p11.2 Deletion
Brief Title: Safety, Tolerability, and Efficacy of Arbaclofen in 16p11.2 Deletion
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Research Associates, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRA16p201
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: 16P11.2 Deletion Syndrome
MeSH Terms: conditions — 16p11.2 Deletion Syndrome | interventions — arbaclofen placarbil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arbaclofen (Experimental): Arbaclofen will be dosed flexibly, with maximum permissible dose depending on age.
  Interventions: Drug: Arbaclofen
- Placebo (Placebo Comparator): The placebo tablet is manufactured to match arbaclofen in shape, size, color, and taste, and will be administered in the same manner as arbaclofen.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Arbaclofen — Arbaclofen tablet
  Other Names: R-baclofen; STX209
  Arms: Arbaclofen
Drug: Placebo oral tablet — Manufactured to match Arbaclofen in size, shape, color and taste
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This Phase 2 study examines the safety, tolerability, and efficacy of arbaclofen in pediatric subjects with 16p11.2 deletion. Male or female subjects aged 5 to 17 years of age will be randomized to receive either placebo or arbaclofen in a double-blind study design. If the subject completes all study requirements through Visit 4 (Close-out Visit), he/she may be eligible for an optional open-label study with arbaclofen.

DETAILED DESCRIPTION:
This study will enroll male or female subjects, aged 5 to 17 years, who have the 16p11.2 bp4-bp5 deletion. Subjects will be randomized to treatment with either placebo or arbaclofen. Subjects and study staff will be blinded to treatment assignment throughout the study. Both placebo and arbaclofen will be administered as orally disintegrating tablets. Dosing will be flexible, with subjects titrating up to the highest tolerated dose, with maximum permissible dose dependent on age. The treatment period is 16 weeks, after which subjects will taper off of study drug. Subjects will be required to attend multiple study visits, and to communicate with the study staff by phone multiple times throughout the study.

The primary efficacy assessment focuses on speech. Secondary and exploratory endpoints assess motor, memory, general cognitive, and other neuropsychological abilities, and brain electrophysiology. The safety evaluations include blood tests, physical exam, and assessment of adverse events.

Subjects who complete study participation through the end of the Withdrawal Period may be eligible to enroll in a subsequent open-label study. Dosing will be flexible, with subjects titrating up to the highest tolerated dose, with maximum permissible dose dependent on age. The treatment period is 16 weeks, after which subjects will taper off arbaclofen.

ELIGIBILITY:
Inclusion Criteria:To be eligible to participate in this study, all of the following criteria must be met:

1. Diagnosis of 16p11.2 BP4-BP5 deletion.
2. Male or female subjects, 5 through 17 years of age, at Screening.
3. Neurodevelopmental disability requiring current educational or other therapeutic support.
4. Any educational, behavioral, other therapeutic, and/or dietary interventions must have been continuous during the 2 months prior to Screening (with the exception of the anti-epileptic drug (AED) 6-month requirement in Inclusion Criterion #5). Subjects and their parent/caregiver/legally authorized representative (LAR) may not electively initiate new, or modify ongoing, interventions for the duration of the study. Typical school vacations are not considered modifications of stable programming.
5. Subjects with a history of seizure disorder must have been seizure-free and on a stable antiepileptic therapy regimen for 6 months OR must have been seizure-free for the 3 years prior to Screening if not currently receiving antiepileptics. If currently receiving treatment with antiepileptics that are typically monitored by serum concentration, serum concentrations of the antiepileptic drugs must be tested and confirmed to be within the therapeutic range at Screening.
6. All medication regimens must be stable for 30 days prior to Screening.
7. Prior to the conduct of any study-specific procedures, the subject must provide assent to participate in the study (if developmentally appropriate), and the parent/caregiver/LAR must provide written informed consent. If the caregiver attending the clinic visits is not the parent or LAR, written consent must also be obtained from the parent or LAR for the subject's participation in the study.
8. The subject's parent/caregiver/LAR must be able to speak and understand English sufficiently to understand the nature of the study and to allow for the completion of all study assessments. The parent/caregiver/LAR should be capable of providing reliable information about the subject's condition, agree to oversee the administration of the study drug, and accompany the subject to all clinic visits. The same parent/caregiver/LAR should accompany the subject to each visit.
9. Negative pregnancy test for females who are 9 years of age or older. Both male and female subjects who are sexually active must agree to consistently use an accepted form of contraception (i.e., surgical sterilization, intrauterine contraceptive device, subcutaneous implant, oral contraceptive, or diaphragm or condom in combination with contraceptive cream/jelly, or abstinence) throughout the trial and for 30 days (females) or 90 days (males) following last study drug administration.

Exclusion Criteria:Subjects are not permitted to enroll in the study if any of the following criteria are met:

1. Subjects with additional known genetic disorder besides 16p11.2 BP4-BP5 deletion.
2. Subjects receiving remote or hybrid schooling at Screening.
3. Subjects with an additional neurologic or psychiatric condition that might confound performance on assessments measures, e.g., significant impairment in hearing or vision, severe motor impairment (e.g., non-ambulatory) from cerebral palsy, birth injury, or other injury, or cleft lip or palate (including submucous cleft).
4. Subjects with any seizures within the previous 6 months; subjects who are not currently receiving antiepileptics AND have had one or more seizures during the 3 years prior to Screening; and subjects who are shown to have non-therapeutic AED levels at Screening.
5. Subjects with any medical or psychiatric condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. This includes, but is not limited to substance use disorders, impairment of renal function, evidence or history of malignancy or any significant hematological, endocrine, cardiovascular, respiratory, hepatic, or gastrointestinal disease.
6. Subjects who plan to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study.
7. Subjects who are currently treated or have been treated with racemic baclofen in the last 30 days.
8. Subjects currently treated with antipsychotic medication(s).
9. Subjects currently treated with more than 2 psychoactive medications, including antiepileptics used as an anti-seizure treatment, but not including sleep aids used on an as-needed basis.
10. Subjects currently treated with drugs having anxiolytic properties, including but not limited to: buspirone and beta-blockers. Benzodiazepines administered on a regular schedule (more than 3x/week) are not permitted. Use of antidepressants may be permitted with approval of the Medical Monitor. Other prohibited and restricted medications are shown in Appendix A.
11. Subjects currently treated with vigabatrin, tiagabine, or riluzole.
12. Subjects taking another investigational drug currently or within the last 30 days.
13. Subjects who are not able or willing to take oral disintegrating tablets.
14. Subjects who have a history of hypersensitivity to racemic baclofen.
15. Subjects who, in the Investigator's opinion, might not be suitable for the study.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-22 (Estimated); Study Completion 2025-03-23 (Estimated)

PRIMARY OUTCOMES:
Goldman-Fristoe Test of Articulation, 3rd edition (GFTA-3), Sounds-in-Words | 12 weeks
  The GFTA-3 is the most widely used, standardized test of articulation for children and adolescents.

SECONDARY OUTCOMES:
Wide Range Assessment of Memory and Learning - 2nd edition (WRAML2) | 12 weeks
  The WRAML2 is a standardized test that measures memory functioning.
Bruininks-Oseretsky Test - 2nd edition (BOT-2), Fine Motor Control and Body Coordination subtests | 12 weeks
  The BOT-2 is an individually administered, comprehensive measure of gross and fine motor skills.
Differential Ability Scale, 2nd edition (DAS-II) | 12 weeks
  The DAS-II is an individually-administered clinical instrument for assessing the cognitive abilities that are important to learning.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wang, MD, Study Director — Clinical Research Associates, LLC
Locations (4):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - New York State Psychiatric Institute (NYSPI), New York, New York
  - Texas Children's Hospital, Houston, Texas
  - University of Washington, Seattle, Washington